CLINICAL TRIAL: NCT04772040
Title: Impact of Omega (ω)-3 Polyunsaturated Fatty Acids (n-3 PUFA) Upon Blood, Muscle and Adipose Tissue Content and Function: Dosing and Washout Study
Brief Title: Impact of Fish Oil Dose on Tissue Content and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Milena Banic, PhD Researcher, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 280280
Record Dates: First submitted 2020-11-04; First posted 2021-02-26 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Aging; Sarcopenia; Muscle Atrophy
Keywords: Omega-3 polyunsaturated fatty acids; Fish oil supplementation; Washout; Dosing strategy
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young loading dose group (Experimental): Participants (18-35) will receive a loading dose of fish oil supplementation during the first 4 weeks of the intervention period of the study. In the last 8 weeks participants will receive a maintenance dose of fish oil supplementation. The total amount of EPA/DHA received throughout the supplementation period will be the same as the old group.
  Interventions: Dietary Supplement: Fish oil supplementation
- Old loading dose group (Experimental): Participants (60y+) will receive a loading dose of fish oil supplementation during the first 4 weeks of the intervention period of the study. In the last 8 weeks participants will receive a maintenance dose of fish oil supplementation. The total amount of EPA/DHA received throughout the supplementation period will be the same as the young group.
  Interventions: Dietary Supplement: Fish oil supplementation
- Young constant dose group (Experimental): Participants (18-35y) will receive a constant dose of fish oil supplementation throughout the intervention period of the study. Total amount of EPA/DHA received throughout the 12 weeks supplementation period will be the same as the loading groups.
  Interventions: Dietary Supplement: Fish oil supplementation
- Old constant dose group (Experimental): Participants (60y+) will receive a constant dose of fish oil supplementation throughout the intervention period of the study. Total amount of EPA/DHA received throughout the 12 weeks supplementation period will be the same as the loading groups.
  Interventions: Dietary Supplement: Fish oil supplementation

INTERVENTIONS:
Dietary Supplement: Fish oil supplementation — Fish oil capsules.

SUMMARY:
In this 5-month study, we will track the incorporation and washout of n-3 PUFA into different tissues following two different dosing strategies in healthy young and older volunteers. All groups will be followed for washout.

Data gathered from this study will be used to establish novel dosing strategies and provide insights into the incorporation of n-3 PUFAs in different tissues and their washout in young and older participants.

DETAILED DESCRIPTION:
Skeletal muscle is crucial for health and accounts for approximately 40% of total body mass. A loss of skeletal muscle mass is seen in the process of ageing, with reductions between 0.2%-0.5% of muscle mass per year starting in the fifth decade. Accelerated loss of muscle and function above a certain threshold is characterized as sarcopenia. Age-related sarcopenia is prevalent in the UK; it is estimated to affect 4.6% men and 7.9% women with an average age of 67 years. Older people have an impaired capacity to increase muscle protein synthesis (MPS) rates in response to protein intake; this is thought to be a key contributor to age-related sarcopenia. Therefore, it is essential to elucidate new strategies to prevent and treat the accelerated loss of muscle mass and function.

Omega (ω)-polyunsaturated fatty acids (n-3 PUFAs) derived from fish oil have possible beneficial effects on health. Evidence suggests potential therapeutic effects of n-3 PUFAs in maintenance/prevention of loss of skeletal muscle mass. N-3 PUFAs probably exert their effects by incorporation into tissue membranes. However, the relation between dose and incorporation into tissue membranes is unclear. Interestingly, a higher dose ingested over 4 weeks seen by McGlory et al. induced similar omega-3 incorporation in the tissue compared to the low doses over 8 weeks studied by Smith et al. If higher doses change tissue composition earlier, then there will be earlier benefits for muscle health and function. Thus, there is a need to examine whether an initial loading dose incorporation into tissues can be sustained by moving to a lower maintenance feeding dose. Furthermore, the exact molecular mechanisms of how n-3 PUFAs act on skeletal muscle are unclear. Several metabolic and molecular responses are affected, but wherein these pathways n-3 PUFAs act remain largely unknown and requires more investigation, with a focus on long-term settings.

This study aims to tackle these problems by executing a 5-month study where we will track the incorporation and washout of n-3 PUFAs into different tissues following two different dosing strategies in healthy young and older volunteers. Data gathered from this study will be used to establish novel dosing strategies and provide insights into the incorporation of n-3 PUFAs in different tissues and their washout in young and older participants. Ultimately, these insights will help targeting, prevention, and treatment of sarcopenia.

Participating in this study requires approximately 30 hours of commitment, of which 12 hours will be spent in the lab.

ELIGIBILITY:
Inclusion Criteria:

* Provide valid informed consent prior to any study procedure
* Males and females 18-35 years of age or 60+ years of age
* BMI between 18-29 kg/m2
* Free of musculoskeletal injuries
* Willing to avoid alcohol in the 48-h period prior to the visits
* Willing to sustain their current diet and lifestyle and not to make conscious changes for the duration of the study
* An omega-3 status of less than 20% seen in whole blood taken during the screening visit.
* Willing to sustain current use of supplementation/anti-depressants or other medication not interfering with the study results.
* Women: not currently pregnant, not intending to become pregnant in the coming 5 months or lactating.
* Women: willing to maintain current use of contraceptives or post-menopausal supplementation if any for the duration of the study.
* Not allergic to fish, shellfish, seaweed, iodine, anesthetics, nickel or chrome.

Exclusion Criteria:

* Smoker
* Adherence to a strict vegan/vegetarian diet
* Treatment for cardiovascular diseases or blood pressure >140/90 mmHg
* Any diseases or medication that cause fat malabsorption (intestine issues such as celiac disease, Crohn's disease,chronic pancreatitis, or cystic fibrosis; liver and biliary disease, diarrhoea, steatorrhea)
* Diabetes or other (metabolic) disease that induce muscle wasting
* Surgery in prior 6 months
* Currently being on FO supplementation
* Current participation in another clinical trial, or in a trial within the past month
* For women: pregnant, intention to get pregnant during the course of the study or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Red blood cell lipid composition | Screening, Baseline (0 weeks), 4 weeks, 6 weeks, 8 weeks, 12 weeks (post intervention), 14 weeks, 16 weeks, 20 weeks (post wash-out)
  Changes in red blood cell membrane lipid composition by collecting venous blood samples.
Skeletal muscle lipid composition | Baseline (0 weeks), 4 weeks, 12 weeks (post-intervention), 20 weeks (post wash-out)
  Changes in skeletal muscle lipid composition by performing a muscle tissue biopsy in the vastus lateralis.
Adipose tissue lipid composition | Baseline (0 weeks), 4 weeks, 12 weeks (post-intervention), 20 weeks (post wash-out)
  Changes in adipose lipid composition by performing an adipose tissue biopsy in the abdominal region.

SECONDARY OUTCOMES:
Skeletal muscle tissue biopsy muscle protein turnover markers | Baseline (0 weeks), 4 weeks, 12 weeks (post-intervention), 20 weeks (post wash-out)
  Secondary outcome from the skeletal muscle biopsy will focus on the measurement of the phosphorylation status of signaling proteins known to regulate protein synthesis and breakdown.
Adipose tissue biopsy inflammation markers | Baseline (0 weeks), 4 weeks, 12 weeks (post-intervention), 20 weeks (post wash-out)
  Secondary outcome from the adipose tissue biopsy will focus on markers involved in inflammation (e.g. NF-kB, IL-6)
Red blood cell lipid mediator markers | Baseline (0 weeks), 4 weeks, 12 weeks (post-intervention), 20 weeks (post wash-out)
  Secondary outcome measures from red blood cells will focus on mediators derived from lipid and changes in lipid mediator synthesis.

OTHER OUTCOMES:
Body composition DEXA scan. | Baseline (0 weeks), 12 weeks (post-intervention), 20 weeks (post wash-out)
  Body composition will be estimated using dual energy X-ray absorptiometry (DEXA) scan.
Subcutaneous fat determination. | Baseline (0 weeks), 12 weeks (post-intervention), 20 weeks (post wash-out)
  Subcutaneous fat will be assessed with the sum of skinfold thicknesses from 8 sites, following the ISAK protocol.
Strength measures | Screening (baseline, 0 weeks), 8 weeks, 16 weeks.
  Muscle strength is determined by performing the handgrip strength test.
Mobility measures | Screening (baseline, 0 weeks), 8 weeks, 16 weeks.
  Muscle mobility is determined by performing the timed-up-and-go test.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Banic, Msc, Principal Investigator — University of Stirling; Nidia Rodriguez-Sanchez, PhD, Study Director — University of Stirling; Stuart Galloway, PhD, Study Director — University of Stirling; Oliver Witard, PhD, Study Director — King's College London; Miriam van Dijk-Ottens, PhD, Study Director — Danone Nutricia Research
Locations (1):
- University of Stirling, Stirling, Stirlingshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No